CLINICAL TRIAL: NCT02757352
Title: A 52-Week Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Ixekizumab (LY2439821) in bDMARD Naive Patients With Nonradiographic Axial Spondyloarthritis
Brief Title: A Study of Ixekizumab (LY2439821) in Participants With Nonradiographic Axial Spondyloarthritis
Acronym: COAST-X
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16180; I1F-MC-RHBX (Other: Eli Lilly and Company); 2015-003938-27 (EudraCT Number)
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Results first posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2019-08-01

CONDITIONS: Axial Spondyloarthritis
Keywords: ankylosing; nonradiographic spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Q2W Ixekizumab (Experimental): Participants received a starting dose of 80 or 160 milligram (mg) of ixekizumab given subcutaneously (SC) at week 0 followed by 80 mg ixekizumab given SC every two weeks (Q2W) to week 52 during the double-blind period.
  Inadequate responders (IR) as determined by investigators could switch to ixekizumab 80 mg Q2W open label between week 16 and 44.
  Interventions: Drug: Ixekizumab
- Q4W Ixekizumab (Experimental): Participants received a starting dose of 80 or 160 mg of ixekizumab given SC at week 0 followed by 80 mg ixekizumab given SC every four weeks (Q4W) to week 52 during the double-blind period.
  Inadequate responders as determined by investigators could switch to ixekizumab 80 mg Q2W open label week 16 and 44.
  Interventions: Drug: Ixekizumab
- Placebo (Placebo Comparator): Participants received placebo as 2 SC injections Q2W to week 52 during double-blind period.
  Inadequate responders as determined by investigators could switch to ixekizumab 80 mg Q2W open label between week 16 and 44.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
  Arms: Q2W Ixekizumab; Q4W Ixekizumab
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of the study drug known as ixekizumab in biologic disease modifying antirheumatic drug (bDMARD) naïve participants with nonradiographic axial spondyloarthritis (nonrad-axSpA).

ELIGIBILITY:
Inclusion Criteria:

* Are ambulatory.
* Diagnosis of nonradiographic axial spondyloarthritis (nr-axSpA) and fulfilling the 2009 Assessment of Spondyloarthritis International Society (ASAS) classification criteria.
* Have a history of back pain ≥3 months with age at onset <45 years.
* Have active nr-axSpA defined as BASDAI ≥4 and total back pain ≥4 on a numeric rating scale (NRS) at screening and baseline.
* Have objective signs of inflammation by presence of sacroiliitis on MRI and/or presence of elevated C-reactive protein (CRP).
* In the past had an inadequate response to at least 2 non-steroidal anti-inflammatory drugs (NSAIDS) for duration of 4 weeks or cannot tolerate NSAIDS.
* If taking NSAIDS be on stable dose for at least 2 weeks prior to randomization.
* Have a history of prior therapy for axSpA for at least 12 weeks prior to screening.

Exclusion Criteria:

* Have radiographic sacroiliitis fulfilling the 1984 modified New York criteria.
* Have received any prior, or are currently receiving treatment with biologics, tumor necrosis factor inhibitors or other immunomodulatory agents.
* Have received a live vaccine within 12 weeks or have had a vaccination with Bacillus Calmette-Guerin (BCG) within the past year.
* Have an ongoing or serious infection within the last 12 weeks or evidence of active tuberculosis.
* Have a compromised immune system.
* Have any other serious and/or uncontrolled diseases.
* Have either a current diagnosis or a recent history of malignant disease.
* Have had major surgery within 8 weeks of baseline, or will require surgery during the study.
* Are pregnant or breastfeeding.
* Have evidence of active anterior uveitis (an acute episode) within the last 42 days prior to baseline randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (103):
- United States (25):
  - Arizona Arthritis Research, PLC, Phoenix, Arizona
  - TriWest Research Assocaites, El Cajon, California
  - Rheumatology Center of San Diego, Escondido, California
  - Care Access Research - Huntington Beach, Huntington Beach, California
  - Desert Medical Advances, Palm Desert, California
  - Inlande Rheumatology Clinical Trials, Upland, California
  - Arthritis Assoc. & Osteoporosis Ctr of Colorado Springs, LLC, Colorado Springs, Colorado
  - Clinical Research Center of CT/NY, Danbury, Connecticut
  - Sarasota Arthritis Center, Sarasota, Florida
  - West Broward Rheumatology Associates, Inc, Tamarac, Florida
  - Marietta Rheumatology, Marietta, Georgia
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - The Arthritis & Diabetes Clinic Inc., Monroe, Louisiana
  - Osteoporosis And Clinical Trial Center, Cumberland, Maryland
  - Osteoporosis And Clinical Trial Center, Hagerstown, Maryland
  - Glacier View Research Institute, Kalispell, Montana
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Weill Cornell Physicians at Brooklyn Heights, Brooklyn, New York
  - Shanahan Rheumatology & Immunotherapy, Raleigh, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Articularis Healthcare Group, INC dba Columbia Arthritis Ctr, Columbia, South Carolina
  - Seattle Rheumatology Associates, P.L.L.C., Seattle, Washington
  - Arthritis Northwest Rheumatology, Spokane, Washington
- Argentina (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Capital Federal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ciudad Autonoma de Buenos Aire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Quilmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, San Miguel de Tucumán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Vienna
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Vienna
- Brazil (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiás
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Juiz de Fora
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Rio de Janeiro
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Québec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, St. John's
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Trois-Rivières
- Czechia (5):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ostrava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pardubice
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Uherské Hradiště
- Finland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Hyvinkää
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Kuopio
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Oulu
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle, Saxony-Anhalt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Bad Doberan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Herne
- Japan (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Bunkyō City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Chūōku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kita-gun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kuwana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Nankoku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nishinomiya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōsaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Sasebo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Suita-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tenri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamagata
- Mexico (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexicali
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mérida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Amsterdam, Netherlands
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Nadarzyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Świdnik
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Puerto Rico (4):
  - Office: Perez-De Jesus, Amarilis, Caguas, PR
  - Ponce School of Medicine CAIMED Center, Ponce, PR
  - Mindful Medical Research, San Juan, PR
  - Latin Clinical Trial Center, Santurce
- Romania (3):
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Constanța
- Russia (6):
  - V.A. Nasonova Research Institute of Rheumatology, Moscow
  - City Clinical Hospital #1, Moscow
  - Ryazan State Medical University/Ryazan Clinical Regional Cardiological Dispensary, Ryazan
  - Clinical Rheumatology Hospital # 25, Saint Petersburg
  - Saratov Regional Clinical Hospital, Saratov
  - Clinical Hospital for Emergency Care, Yaroslavl
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Reveille JD, Rudwaleit M, Rahman P, Maldonado-Cocco JA, Magrey M, Bolce R, Ng KJ, Gibble TH, Lisse J, Park SY, Kronbergs A, Navarro-Compan V. Does HLA-B27 Status Influence Ixekizumab Efficacy in Axial Spondyloarthritis? Results From the COAST-V, COAST-W, and COAST-X Trials. Rheumatol Ther. 2026 Feb;13(1):279-291. doi: 10.1007/s40744-025-00810-5. Epub 2025 Dec 19. PMID 41417207
- [Derived] Navarro-Compan V, Reveille JD, Rahman P, Maldonado-Cocco JA, Magrey M, Bolce R, Panni T, Kronbergs A, Rudwaleit M. Ixekizumab Improves Signs, Symptoms, and Quality of Life in Patients with Axial Spondyloarthritis Irrespective of Symptom Duration. Adv Ther. 2025 Sep;42(9):4706-4716. doi: 10.1007/s12325-025-03305-5. Epub 2025 Jul 22. PMID 40694276
- [Derived] Maksymowych WP, Baraliakos X, Lambert RG, Landewe R, Sandoval D, Carlier H, Lisse J, Li X, Hojnik M, Ostergaard M. Effects of ixekizumab treatment on structural changes in the sacroiliac joint: MRI assessments at 16 weeks in patients with non-radiographic axial spondyloarthritis. Lancet Rheumatol. 2022 Sep;4(9):e626-e634. doi: 10.1016/S2665-9913(22)00185-0. Epub 2022 Aug 9. PMID 38288892
- [Derived] Deodhar A, Poddubnyy D, Rahman P, Ermann J, Tomita T, Bolce R, Leage SL, Kronbergs A, Johnson C, Araujo J, Leung A, van der Heijde D. Long-Term Safety and Efficacy of Ixekizumab in Patients With Axial Spondyloarthritis: 3-year Data From the COAST Program. J Rheumatol. 2023 Aug;50(8):1020-1028. doi: 10.3899/jrheum.221022. Epub 2023 Feb 15. PMID 36792107
- [Derived] Ortolan A, Ramiro S, Ramonda R, van der Heijde D. External validation of the alternative Ankylosing Spondylitis Disease Activity Score in three randomized clinical trials of ixekizumab. Rheumatology (Oxford). 2023 Jun 1;62(6):2257-2261. doi: 10.1093/rheumatology/keac618. PMID 36282526
- [Derived] van der Horst-Bruinsma IE, de Vlam K, Walsh JA, Bolce R, Hunter T, Sandoval D, Zhu D, Geneus V, Soriano ER, Magrey M. Baseline Characteristics and Treatment Response to Ixekizumab Categorised by Sex in Radiographic and Non-radiographic Axial Spondylarthritis Through 52 Weeks: Data from Three Phase III Randomised Controlled Trials. Adv Ther. 2022 Jun;39(6):2806-2819. doi: 10.1007/s12325-022-02132-2. Epub 2022 Apr 16. PMID 35429281
- [Derived] Deodhar A, Mease P, Marzo-Ortega H, Hunter T, Sandoval D, Kronbergs A, Lauzon S, Leung A, Navarro-Compan V. Ixekizumab improves sleep and work productivity in patients with non-radiographic axial spondyloarthritis: results from the COAST-X trial at 52 weeks. BMC Rheumatol. 2021 Sep 25;5(1):50. doi: 10.1186/s41927-021-00218-y. PMID 34560906
- [Derived] Deodhar A, Mease P, Rahman P, Navarro-Compan V, Marzo-Ortega H, Hunter T, Sandoval D, Kronbergs A, Leon L, Shan M, Leung A, De Vlam K, Strand V. Ixekizumab Improves Patient-Reported Outcomes in Non-Radiographic Axial Spondyloarthritis: Results from the Coast-X Trial. Rheumatol Ther. 2021 Mar;8(1):135-150. doi: 10.1007/s40744-020-00254-z. Epub 2020 Dec 7. PMID 33284423
- [Derived] Walsh JA, Magrey MN, Baraliakos X, Inui K, Weng MY, Lubrano E, van der Heijde D, Boonen A, Gensler LS, Strand V, Braun J, Hunter T, Li X, Zhu B, Leon L, Calderon DMS, Kiltz U. Improvement of Functioning and Health With Ixekizumab in the Treatment of Active Nonradiographic Axial Spondyloarthritis in a 52-Week, Randomized, Controlled Trial. Arthritis Care Res (Hoboken). 2022 Mar;74(3):451-460. doi: 10.1002/acr.24482. Epub 2022 Jan 26. PMID 33044756
- [Derived] Deodhar A, van der Heijde D, Gensler LS, Kim TH, Maksymowych WP, Ostergaard M, Poddubnyy D, Marzo-Ortega H, Bessette L, Tomita T, Leung A, Hojnik M, Gallo G, Li X, Adams D, Carlier H, Sieper J; COAST-X Study Group. Ixekizumab for patients with non-radiographic axial spondyloarthritis (COAST-X): a randomised, placebo-controlled trial. Lancet. 2020 Jan 4;395(10217):53-64. doi: 10.1016/S0140-6736(19)32971-X. Epub 2019 Dec 5. PMID 31813637
- See also: Click here for more information about this study: A Study of Ixekizumab (LY2439821) in Participants With Nonradiographic Axial Spondyloarthritis (COAST-X) — http://www.lillytrialguide.com/en-US/studies/nonradiographic-axial%20spondyloarthritis/RHBX#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study has 3 periods: Period 1 - Screening; Period 2 - A Double-Blind Treatment Period (Weeks 0 Up to 52); (Inadequate Responders [IR] Week 16-52) followed by a Follow-Up Period (Up to 24 Weeks after last visit)
Pre-assignment Details: Participants who completed study were eligible to enroll into a long-term study (Study I1F-MC-RHBY [RHBY]) for up to 2 additional years. Participants that do not enroll into study RHBY will complete the Post-Treatment Follow-Up Period.
Groups:
- Placebo Double-Blind Period: Participants received placebo (PBO) as 2 subcutaneous (SC) injections every two weeks (Q2W) to week 52.
- Ixekizumab 80 mg Q4W (IxeQ4W) Double-Blind Period: Participants received a starting dose of 80 or 160 milligram (mg) of ixekizumab given subcutaneously (SC) at week 0 followed by 80 mg ixekizumab given SC every four weeks (Q4W) to week 52.
- Ixekizumab 80 mg Q2W (IxeQ2W) Double-Blind Period: Participants received a starting dose of 80 or 160 mg of ixekizumab given SC at week 0 followed by 80 mg ixekizumab given SC (Q2W) to week 52.
- PBO IR/Ixe80Q2W-Open Label: Participants who received placebo in double blind period and were inadequate responders as determined by investigators switched to ixekizumab 80 mg Q2W open label.
- Ixekizumab 80 mg Q4W IR (Ixe80Q4WIR)/Ixe80Q2W-Open Label: Participants who received ixekizumab 80 mg Q4W in double blind period and were inadequate responders as determined by investigators switched to ixekizumab 80 mg Q2W open label.
- Ixekizumab 80 mg Q2W IR (Ixe80Q2WIR)/Ixe80Q2W-Open Label: Participants who received ixekizumab 80 mg Q2W in double blind period and were inadequate responders as determined by investigators continued on the same regimen of ixekizumab 80 mg Q2W open label.
- Placebo Post Treatment Follow-Up Period: Participants discontinued the study early and entered the post-treatment follow-up period. Participants received placebo immediately prior to entering the post-treatment follow-up period.
- Ixekizumab 80 mg Q4W Post Treatment Follow-Up Period: Participants discontinued the study early and entered the post-treatment follow-up period. Participants received ixekizumab 80 mg Q4W immediately prior to entering the post-treatment follow-up period.
- Ixekizumab 80 mg Q2W Post Treatment Follow-Up Period: Participants discontinued the study early and entered the post-treatment follow-up period. Participants received ixekizumab 80 mg Q2W immediately prior to entering the post-treatment follow-up period
- Other Biologic Treatment Group: Participants who discontinued study treatment and were on other biologic therapy prior to entering follow-up period.
Period: Double-Blind Period (Week 0 - Week 16)
Arm/Group | Placebo Double-Blind Period | Ixekizumab 80 mg Q4W (IxeQ4W) Double-Blind Period | Ixekizumab 80 mg Q2W (IxeQ2W) Double-Blind Period | PBO IR/Ixe80Q2W-Open Label | Ixekizumab 80 mg Q4W IR (Ixe80Q4WIR)/Ixe80Q2W-Open Label | Ixekizumab 80 mg Q2W IR (Ixe80Q2WIR)/Ixe80Q2W-Open Label | Placebo Post Treatment Follow-Up Period | Ixekizumab 80 mg Q4W Post Treatment Follow-Up Period | Ixekizumab 80 mg Q2W Post Treatment Follow-Up Period | Other Biologic Treatment Group
Started | 105 | 96 | 102 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 104 | 96 | 102 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 97 | 95 | 98 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-Blind Period (Week 16 - Week 52)
Arm/Group | Placebo Double-Blind Period | Ixekizumab 80 mg Q4W (IxeQ4W) Double-Blind Period | Ixekizumab 80 mg Q2W (IxeQ2W) Double-Blind Period | PBO IR/Ixe80Q2W-Open Label | Ixekizumab 80 mg Q4W IR (Ixe80Q4WIR)/Ixe80Q2W-Open Label | Ixekizumab 80 mg Q2W IR (Ixe80Q2WIR)/Ixe80Q2W-Open Label | Placebo Post Treatment Follow-Up Period | Ixekizumab 80 mg Q4W Post Treatment Follow-Up Period | Ixekizumab 80 mg Q2W Post Treatment Follow-Up Period | Other Biologic Treatment Group
Started | 97 | 95 | 98 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 34 | 52 | 52 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 63 | 43 | 46 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Classified as Inadequate Responders (IR) | 62 | 40 | 42 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: IR-Open Label Period (Week 16 - Week 52)
Arm/Group | Placebo Double-Blind Period | Ixekizumab 80 mg Q4W (IxeQ4W) Double-Blind Period | Ixekizumab 80 mg Q2W (IxeQ2W) Double-Blind Period | PBO IR/Ixe80Q2W-Open Label | Ixekizumab 80 mg Q4W IR (Ixe80Q4WIR)/Ixe80Q2W-Open Label | Ixekizumab 80 mg Q2W IR (Ixe80Q2WIR)/Ixe80Q2W-Open Label | Placebo Post Treatment Follow-Up Period | Ixekizumab 80 mg Q4W Post Treatment Follow-Up Period | Ixekizumab 80 mg Q2W Post Treatment Follow-Up Period | Other Biologic Treatment Group
Started | 0 (Participants continued with original assigned treatment without switching to open label ixeQ2W.) | 0 (Participants continued with original assigned treatment without switching to open label ixeQ2W.) | 0 (Participants continued with original assigned treatment without switching to open label ixeQ2W.) | 62 (IR based on the investigator's opinion switched to ixekizumab open label 80 mg Q2W.) | 40 (IR based on the investigator's opinion switched to ixekizumab open label 80 mg Q2W.) | 42 (IR based on the investigator's opinion switched to ixekizumab open label 80 mg Q2W.) | 0 | 0 | 0 | 0
Initiated Other Biologic Rescue | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 55 | 37 | 35 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 7 | 3 | 7 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 2 | 1 | 4 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Period: Follow-Up Period
Arm/Group | Placebo Double-Blind Period | Ixekizumab 80 mg Q4W (IxeQ4W) Double-Blind Period | Ixekizumab 80 mg Q2W (IxeQ2W) Double-Blind Period | PBO IR/Ixe80Q2W-Open Label | Ixekizumab 80 mg Q4W IR (Ixe80Q4WIR)/Ixe80Q2W-Open Label | Ixekizumab 80 mg Q2W IR (Ixe80Q2WIR)/Ixe80Q2W-Open Label | Placebo Post Treatment Follow-Up Period | Ixekizumab 80 mg Q4W Post Treatment Follow-Up Period | Ixekizumab 80 mg Q2W Post Treatment Follow-Up Period | Other Biologic Treatment Group
Started | 0 | 0 | 0 | 0 (Participants who completed the study were eligible to enroll in RHBY or enter follow up period.) | 0 (Participants who completed the study were eligible to enroll in RHBY or enter follow up period.) | 0 (Participants who completed the study were eligible to enroll in RHBY or enter follow up period.) | 3 (Participants who completed the study were eligible to enroll in RHBY or enter follow up period.) | 5 (Participants who completed the study were eligible to enroll in RHBY or enter follow up period.) | 28 (Participants who completed the study were eligible to enroll in RHBY or enter follow up period.) | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 18 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 10 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo: Participants received placebo as 2 SC injections Q2W to week 52.
- Ixekizumab 80 mg Q4W: Participants received a starting dose of 80 or 160 mg of ixekizumab given SC at week 0 followed by 80 mg ixekizumab given SC every four weeks (Q4W) to week 52.
- Ixekizumab 80 mg Q2W: Participants received a starting dose of 80 or 160 mg of ixekizumab given SC at week 0 followed by 80 mg ixekizumab given SC every two weeks (Q2W) to week 52.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W | Total
Number analyzed (Participants) | 105 | 96 | 102 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Participants who had evaluable data for age were reported due to 1 participant that did not receive study drug.
  years
    number analyzed (Participants) | 104 | 96 | 102 | 302
    (all) | 39.9 (12.36) | 40.9 (14.47) | 40.0 (12.01) | 40.3 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 46 | 53 | 160
  Male | 44 | 50 | 49 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 24 | 31 | 80
  Not Hispanic or Latino | 68 | 57 | 63 | 188
  Unknown or Not Reported | 12 | 15 | 8 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 2 | 3 | 13
  Asian | 17 | 13 | 11 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 76 | 80 | 83 | 239
  More than one race | 3 | 1 | 5 | 9
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 8 | 6 | 9 | 23
  Romania | 5 | 1 | 4 | 10
  United States | 10 | 9 | 9 | 28
  Czechia | 15 | 16 | 13 | 44
  Japan | 6 | 5 | 5 | 16
  Russia | 12 | 7 | 8 | 27
  Canada | 1 | 3 | 2 | 6
  Austria | 0 | 1 | 2 | 3
  South Korea | 9 | 7 | 6 | 22
  Netherlands | 0 | 0 | 1 | 1
  Finland | 4 | 3 | 3 | 10
  Brazil | 0 | 1 | 2 | 3
  Poland | 19 | 18 | 20 | 57
  Mexico | 14 | 13 | 15 | 42
  Germany | 2 | 6 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an Assessment of Spondyloarthritis International Society 40 (ASAS40) Response
Description: ASAS40 is defined as a greater than or equal to (≥)40% improvement and an absolute improvement from baseline of ≥2 units (ranges 0 to 10) in at least 3 of the 4 domains (Patient Global, Spinal Pain, Function, and Inflammation), without any worsening in the remaining domain. 1) Patient Global: How active was your spondylitis during the last week? score ranges 0 (not active) to 10 (very active). 2) Spinal Pain: How much spinal pain due to Ankylosing spondylitis? score ranges 0 (no pain) to 10 (severe pain). 3) Bath Ankylosing Spondylitis Functional Index: Participant is asked to rate the difficulty associated with 10 individual basic functional activities. Responses were captured using numeric rating scale (NRS) (ranges 0 to 10) with a higher score of worse function. 4) Inflammation based on mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) question 5 and 6 (mean of intensity, duration of stiffness). Score ranges (0 (non) to 10 (very severe).
Time Frame: Week 16
Population: All randomized participants. For inadequate responders who were treated with open label ixekizumab 80 mg Q2W, only data up to the time of initiation of open label of ixekizumab 80 mg Q2W were included. Missing data was imputed using the nonresponder imputation (NRI) method.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
percentage of participants | 19.0 | 35.4 | 40.2
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.009, Regression, Logistic; Odds Ratio (OR) = 2.36, 95% CI 2-sided [1.23 to 4.51]
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.78, 95% CI 2-sided [1.48 to 5.25]

2. Primary Outcome: Percentage of Participants Achieving an ASAS40 Response
Description: as for outcome 1
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
percentage of participants | 13.3 | 30.2 | 31.4
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 2.82, 95% CI 2-sided [1.38 to 5.77]
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.004, Regression, Logistic; Odds Ratio (OR) = 2.85, 95% CI 2-sided [1.40 to 5.77]

3. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS)
Description: ASDAS is a composite index to assess disease activity in axial spondyloarthritis (axSpA). ASDAS parameters used with (C-reactive protein [CRP] as acute phase reactant) are: 1) Total back pain 2) Patient global 3) Peripheral pain/swelling, duration of morning stiffness 4) CRP in mg/L: ASDAScrp is calculated with the equation: 0.121 × total back pain + 0.110×patient global + 0.073 × peripheral pain/swelling + 0.058 × duration of morning stiffness + 0.579 × Ln(CRP+1). CRP is in milligram/liter (mg/L), the range of other variables is from 0 to 10. Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher scores indicated higher disease activity. Ln represents the natural logarithm. Least squares mean (LS Mean) was derived from mixed models repeated measure analysis (MMRM) with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants. For inadequate responders who were treated with open label ixekizumab 80 mg Q2W, only data up to the time of initiation of open label of ixekizumab 80 mg Q2W were included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
score on a scale | -0.58 (0.095) | -1.12 (0.097) | -1.26 (0.095)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.54, 95% CI 2-sided [-0.81 to -0.28], Standard Error of Mean 0.136
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.68, 95% CI 2-sided [-0.94 to -0.41], Standard Error of Mean 0.134

4. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS)
Description: ASDAS is a composite index to assess disease activity in axSpA. ASDAS parameters used (with CRP as acute phase reactant) are: 1 )Total back pain 2) Patient global 3) Peripheral pain/swelling 4) Duration of morning stiffness 5) CRP in mg/L: ASDAScrp is calculated with the following equation: 0.121 × total back pain + 0.110 × patient global + 0.073 × peripheral pain/swelling + 0.058 × duration of morning stiffness + 0.579 × Ln(CRP+1). CRP is in milligram/liter (mg/L), the range of other variables is from 0 to 10. Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher scores indicated higher disease activity. Ln represents the natural logarithm. LS Mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
score on a scale | -0.78 (0.136) | -1.39 (0.116) | -1.47 (0.116)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.61, 95% CI 2-sided [-0.96 to -0.26], Standard Error of Mean 0.179
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.69, 95% CI 2-sided [-1.05 to -0.34], Standard Error of Mean 0.178

5. Secondary Outcome: Number of Participants Without Clinically Meaningful Changes in Background Therapy
Description: Number of participants without changes in background therapy while on originally randomized treatment.
Time Frame: Baseline through Week 52
Population: All randomized participants. Additional analysis not performed due to small number of participants with changes in background therapy and complete overlap with switch to open-label ixekizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
Participants | 98 | 90 | 100

6. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score
Description: The SF-36 is a 36-item patient-administered measure designed to be a short, multipurpose assessment of health in the areas of physical functioning, role - physical, role - emotional, bodily pain, vitality, social functioning, mental health, and general health. The Physical Component Summary score ranges from 0 to 100; higher scores indicate better levels of function and/or better health. LS Mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
score on a scale | 5.2103 (0.7999) | 8.0612 (0.8129) | 7.9600 (0.8023)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.013, Mixed Models Analysis; LS Mean Difference = 2.8509, 95% CI 2-sided [0.6092 to 5.0926], Standard Error of Mean 1.1390
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.015, Mixed Models Analysis; LS Mean Difference = 2.7497, 95% CI 2-sided [0.5299 to 4.9694], Standard Error of Mean 1.1278

7. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score
Description: The medical outcomes study 36-item short-form health survey (SF-36) SF-36 PCS are summarized using the t-scores. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. LS Mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
score on a scale | 4.7210 (1.2459) | 8.9211 (1.0783) | 9.3291 (1.0810)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.012, Mixed Models Analysis; LS Mean Difference = 4.2001, 95% CI 2-sided [0.9525 to 7.4477], Standard Error of Mean 1.6467
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.006, Mixed Models Analysis; LS Mean Difference = 4.6081, 95% CI 2-sided [1.3629 to 7.8533], Standard Error of Mean 1.6455

8. Secondary Outcome: Percentage of Participants Achieving ASDAS Low Disease Activity
Description: ASDAS is a composite index to assess disease activity in axSpA. ASDAS low disease activity is defined as a score of <2.1. The parameters used for the ASDAS (with CRP as acute phase reactant) are total back pain, patient global, peripheral pain/swelling, duration of morning stiffness and CRP in mg/L. The ASDAScrp is calculated with the following equation: 0.121×total back pain+0.110×patient global+0.073×peripheral pain/swelling+0.058×duration of morning stiffness+0.579×Ln(CRP+1). CRP is in mg/liter, the range of other variables is from 0(normal) to 10(very severe); Ln represents the natural logarithm). Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher the score worse the disease activity.
Time Frame: Week 16
Population: All randomized participants with baseline ASDAS <2.1. For inadequate responders who were treated with open label ixekizumab 80 mg Q2W, only data up to the time of initiation of open label of ixekizumab 80 mg Q2W were included. Missing data was imputed using the NRI method.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 94 | 102
percentage of participants | 12.4 | 27.7 | 32.4
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 2.73, 95% CI 2-sided [1.30 to 5.76]
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.43, 95% CI 2-sided [1.66 to 7.08]

9. Secondary Outcome: Percentage of Participants Achieving ASDAS Low Disease Activity
Description: as for outcome 8
Time Frame: Week 52
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 94 | 102
percentage of participants | 8.6 | 29.8 | 27.5
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.58, 95% CI 2-sided [2.02 to 10.41]
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.99, 95% CI 2-sided [1.76 to 9.05]

10. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: The BASDAI is a participant-reported assessment consisting of 6 questions that relate to 5 major symptoms relevant to axial spondyloarthritis (axSpA): 1) Fatigue, 2) Spinal pain, 3) Peripheral arthritis, 4) Enthesitis, 5) Intensity, and 6) Duration of morning stiffness. Participants need to score each item with a score from 0 to 10 (NRS). Total score is obtained from the average of symptom scores ranging 0 (no problem) to 10 (worst problem), with a higher score indicating more severe AS symptom. LS mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
score on a scale | -1.51 (0.216) | -2.18 (0.220) | -2.52 (0.217)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.031, Mixed Models Analysis; LS Means Square Difference = -0.67, 95% CI 2-sided [-1.28 to -0.06], Standard Error of Mean 0.308
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.001, Mixed Models Analysis; LS Mean Difference = -1.01, 95% CI 2-sided [-1.61 to -0.41], Standard Error of Mean 0.305

11. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: as for outcome 10
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
score on a scale | -1.76 (0.305) | -2.89 (0.266) | -3.04 (0.266)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.006, Mixed Models Analysis; LS Mean Difference = -1.13, 95% CI 2-sided [-1.92 to -0.33], Standard Error of Mean 0.404
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.002, Mixed Models Analysis; LS Mean Difference = -1.29, 95% CI 2-sided [-2.08 to -0.49], Standard Error of Mean 0.404

12. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) of the Sacroiliac Joint (SIJ) Spondyloarthritis Research Consortium of Canada (SPARCC) Score
Description: Both left and right SIJ are scored for bone marrow edema. Each side has 6 slices and each slice has 6 scoring units, and each scoring unit has a score of 0 or 1. Total SIJ SPARCC scores can range from 0 to 72 with higher scores reflecting worse disease. LS Mean was derived from ANCOVA model with treatment, geographic region, screening MRI/CRP status and baseline value as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and Week 16 SPARCC score. For inadequate responders who were treated with open label ixekizumab 80 mg Q2W, only data up to the time of initiation of open label of ixekizumab 80 mg Q2W were included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 90 | 85 | 92
score on a scale | -0.31 (0.539) | -3.38 (0.549) | -4.52 (0.530)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -3.07, 95% CI 2-sided [-4.58 to -1.57], Standard Error of Mean 0.764
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = -4.20, 95% CI 2-sided [-5.68 to -2.72], Standard Error of Mean 0.751

13. Secondary Outcome: Change From Baseline in SPARCC Enthesitis Score
Description: The SPARCC enthesitis is an index used to measure the severity of enthesitis. The SPARCC assesses 16 sites for enthesitis using a score of "0" for no activity or "1" for activity. Sites assessed include Medial epicondyle (left/right [L/R]), Lateral epicondyle (L/R), Supraspinatus insertion into greater tuberosity of humerus (L/R), Greater trochanter (L/R), Quadriceps insertion into superior border of patella (L/R), Patellar ligament insertion into inferior pole of patella or tibial tubercle (L/R), Achilles tendon insertion into calcaneum (L/R), and Plantar fascia insertion into calcaneum (L/R). The SPARCC is the sum of all site scores (range 0 to 16). Higher scores indicate more severe enthesitis. LS Mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status, baseline value visit, baseline value-by-visit and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: All randomized participants with a baseline SPARCC score >0. For inadequate responders who were treated with open label ixekizumab 80 mg Q2W, only data up to the time of initiation of open label of ixekizumab 80 mg Q2W were included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 86 | 65 | 74
score on a scale | -2.87 (0.447) | -2.99 (0.427) | -3.14 (0.407)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.849, Mixed Models Analysis; LS Mean Difference = -0.12, 95% CI 2-sided [-1.35 to 1.11], Standard Error of Mean 0.621
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.648, Mixed Models Analysis; LS Mean Difference = -0.28, 95% CI 2-sided [-1.48 to 0.93], Standard Error of Mean 0.608

14. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: BASFI is a participant-reported assessment that establishes a participant's functional baseline and subsequent response to treatment. Participants were asked to rate the difficulty associated with 10 individual basic functional activities. Participant responded to each question using a NRS scale (range 0 to 10), with a higher score indicating worse functioning. The participant's final BASFI score is the mean of the 10 item scores with the minimum value of 0 and a possible maximum value of 10, with a higher score indicating worse function. LS Mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
score on a scale | -1.57 (0.333) | -2.63 (0.292) | -2.75 (0.291)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.018, Mixed Models Analysis; LS Mean Difference = -1.06, 95% CI 2-sided [-1.93 to -0.18], Standard Error of Mean 0.443
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.008, Mixed Models Analysis; LS Mean Difference = -1.18, 95% CI 2-sided [-2.05 to -0.31], Standard Error of Mean 0.442

15. Secondary Outcome: Percentage of Participants Achieving ASDAS Inactive Disease
Description: ASDAS is a composite index to assess disease activity in axSpA. ASDAS Inactive Disease is defined as a score of less than (<)1.3. The parameters used for the ASDAS (with CRP as acute phase reactant) are total back pain, patient global, peripheral pain/swelling, duration of morning stiffness and CRP in mg/L. The ASDAScrp is calculated with the following equation: 0.121×total back pain+0.110×patient global+0.073×peripheral pain/swelling+0.058×duration of morning stiffness+0.579×Ln(CRP+1). (CRP is in mg/liter, the range of other variables is from 0(normal) to 10(very severe); Ln represents the natural logarithm). Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher the score worse the disease activity.
Time Frame: Week 52
Population: All randomized participants. For inadequate responders who were treated with open label ixekizumab 80 mg Q2W, only data up to the time of initiation of open label of ixekizumab 80 mg Q2W were included. Missing data was imputed using the NRI method.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
percentage of participants | 2.9 | 13.5 | 10.8
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.0011, Regression, Logistic; Odds Ratio (OR) = 5.33, 96% CI 2-sided [1.47 to 19.40]
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.031, Regression, Logistic; Odds Ratio (OR) = 4.22, 95% CI 2-sided [1.14 to 15.66]

16. Secondary Outcome: Change From Baseline in the Measure of High Sensitivity C-Reactive Protein (CRP)
Description: High-sensitivity C-reactive protein (hs-CRP) was the measure of acute phase reactant and was measured with a high sensitivity assay at the central laboratory to help assess the effect of ixekizumab on disease activity. LS Mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: milligram/liter (mg/L)
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
milligram/liter (mg/L) | -4.804 (2.0370) | -8.611 (2.0028) | -7.547 (1.9654)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.183, Mixed Models Analysis; LS Mean Difference = -3.807, 95% CI 2-sided [-9.418 to 1.804], Standard Error of Mean 2.8507
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.331, Mixed Models Analysis; LS Mean Difference = -2.743, 95% CI 2-sided [-8.294 to 2.807], Standard Error of Mean 2.8202

17. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI)
Description: Bath Ankylosing Spondylitis Metrology Index (BASMI) is a combined index comprising the following 5 clinical measurements of spinal mobility in participants with axSpA: 1) Lateral spinal flexion 2) Tragus-to-wall distance 3) Lumbar flexion (modified Schrober) 4) Maximal intermalleolar distance, and 5) Cervical rotation. The BASMI includes these 5 measurements that were each scaled to a score of 0 to 10 depending on the result of the assessment (BASMI linear function). The average score of the 5 assessments gives the BASMI linear result. LS Mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
score on a scale | -0.17 (0.112) | -0.56 (0.097) | -0.48 (0.097)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.008, Mixed Models Analysis; LS Mean Difference = -0.40, 95% CI 2-sided [-0.69 to -0.10], Standard Error of Mean 0.148
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.038, Mixed Models Analysis; LS Mean Difference = -0.31, 95% CI 2-sided [-0.60 to -0.02], Standard Error of Mean 0.148

18. Secondary Outcome: Change From Baseline in Chest Expansion
Description: While participants have their hands resting on or behind the head, the assessor has measured the chest's encircled length by centimeter at the fourth intercostal level anteriorly. The difference between maximal inspiration and expiration in centimeters was recorded. Two tries were recorded. The better measurement (larger difference) of 2 tries (in centimeters) was used for analyses. LS Mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: centimeter (cm)
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
centimeter (cm) | 0.57 (0.253) | 0.62 (0.206) | 0.91 (0.209)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.871, Mixed Models Analysis; LS Mean Difference = 0.05, 95% CI 2-sided [-0.59 to 0.70], Standard Error of Mean 0.325
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.295, Mixed Models Analysis; LS Mean Difference = 0.34, 95% CI 2-sided [-0.30 to 0.99], Standard Error of Mean 0.327

19. Secondary Outcome: Change From Baseline in Occiput to Wall Distance
Description: The participant is to make a maximum effort to touch the head against the wall when standing with heels and back against the wall (occiput). Then the distance from occiput to wall is measured. Two tries will be recorded. The better (smaller) measurement of 2 tries (in centimeters) will be used for analyses. LS Mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
cm | 0.04 (0.312) | -0.42 (0.257) | -0.73 (0.259)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.257, Mixed Models Analysis; LS Mean Difference = -0.46, 95% CI 2-sided [-1.26 to 0.34], Standard Error of Mean 0.406
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.057, Mixed Models Analysis; LS Mean Difference = -0.77, 95% CI 2-sided [-1.56 to 0.02], Standard Error of Mean 0.402

20. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES)
Description: Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) is an index used to measure the severity of enthesitis. The MASES assesses 13 sites for enthesitis using a score of "0" for no activity or "1" for activity. Sites assessed included costochondral 1 (right/left [R/L]), costochondral 7 (R/L), spinal iliaca anterior superior (R/L), crista iliaca (R/L), spina iliaca posterior (R/L), processus spinosus L5, and achilles tendon proximal insertion (R/L). The MASES is the sum of all site scores (range 0 to 13); higher scores indicate more severe enthesitis. LS mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: All randomized participants with baseline Mases score > 0. For inadequate responders who were treated with open label ixekizumab 80 mg Q2W, only data up to the time of initiation of open label of ixekizumab 80 mg Q2W were included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
score on a scale | -2.34 (0.361) | -3.21 (0.342) | -3.19 (0.336)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.082, Mixed Models Analysis; LS Mean Difference = -0.87, 95% CI 2-sided [-1.85 to 0.11], Standard Error of Mean 0.496
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.088, Mixed Models Analysis; LS Mean Difference = -0.85, 95% CI 2-sided [-1.82 to 0.13], Standard Error of Mean 0.493

21. Secondary Outcome: Change From Baseline in Severity of Peripheral Arthritis by Tender (TJC) and Swollen Joint Count (SJC) Scores of 44 Joints
Description: The number of tender and painful joints was determined by examination of 46 joints (23 joints on each side of the participants body). The 46 joints are assessed and classified as tender or not tender. Sum of all joints checked to be tender/painful divided by number of evaluable joints which is multiplied by 46 to obtain TJC score. The scores ranges from 0 (no tender/painful joints) to 46 (all joints tender/painful). Swollen joint count SJC was determined by examination of 44 joints (22 joints on each side of the participants body). The joints are classified as swollen or not swollen. Sum of all joints checked to be swollen divided by number of evaluable joints which is multiplied by 44 to obtain SJC score. Score ranges from 0 (not swollen) to 44 (all joints swollen). LS mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status and baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: All randomized participants with baseline TJC>0 for the TJC analysis. All randomized participants with baseline SJC>0 for the SJC analysis. For inadequate responders who were treated with open label ixekizumab 80 mg Q2W, only data up to the time of initiation of open label of ixekizumab 80 mg Q2W were included.
Measure: Least Squares Mean (Standard Error); unit: joint counts
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
joint counts
  TJC: number analyzed (Participants) | 83 | 70 | 86
  TJC | -0.59 (1.039) | -2.38 (0.993) | -4.12 (0.916)
  SJC: number analyzed (Participants) | 50 | 51 | 57
  SJC | -3.66 (0.261) | -4.63 (0.237) | -4.41 (0.228)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; TJC; Test type: Superiority; p = 0.219, Mixed Models Analysis; LS Mean Difference = -1.79, 95% CI 2-sided [-4.66 to 1.09], Standard Error of Mean 1.442
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; TJC; Test type: Superiority; p = 0.013, Mixed Models Analysis; LS Mean Difference = -3.53, 95% CI 2-sided [-6.30 to -0.76], Standard Error of Mean 1.388
Statistical Analysis 3: Comparison: Placebo vs Ixekizumab 80 mg Q4W; SJC; Test type: Superiority; p = 0.009, Mixed Models Analysis; LS Mean Difference = -0.97, 95% CI 2-sided [-1.68 to -0.26], Standard Error of Mean 0.355
Statistical Analysis 4: Comparison: Placebo vs Ixekizumab 80 mg Q2W; SJC; Test type: Superiority; p = 0.034, Mixed Models Analysis; LS Mean Difference = -0.76, 95% CI 2-sided [-1.46 to -0.06], Standard Error of Mean 0.348

22. Secondary Outcome: Number of Participants With Anterior Uveitis
Description: Number of participants with anterior uveitis. Anterior uveitis is an inflammation of the middle layer of the eye which includes the iris (colored part of the eye) and the adjacent tissue, known as the ciliary body.
Time Frame: Baseline through Week 52
Population: All randomized participants regardless of history of anterior uveitis. For inadequate responders who were treated with open label ixekizumab 80 mg Q2W, only data up to the time of initiation of open label of ixekizumab 80 mg Q2W were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
Participants | 2 | 1 | 2

23. Secondary Outcome: Change From Baseline in the Fatigue Numeric Rating Scale (NRS) Score
Description: The Fatigue Severity NRS is a participant-administered, single-item, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no fatigue" and 10 representing "as bad as you can imagine". Participants rate their fatigue (feeling tired or worn out) by circling the one number that describes their worst level of fatigue during the previous 24 hours. LS Mean was derived from MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
score on a scale | -2.1 (0.38) | -2.6 (0.32) | -2.7 (0.32)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.325, Mixed Models Analysis; LS Mean Difference = -0.5, 95% CI 2-sided [-1.5 to 0.5], Standard Error of Mean 0.50
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.206, Mixed Models Analysis; LS Mean Difference = -0.6, 95% CI 2-sided [-1.6 to 0.4], Standard Error of Mean 0.50

24. Secondary Outcome: Change From Baseline in ASAS Health Index (ASAS HI)
Description: ASAS-HI is a disease-specific health-index instrument designed to assess the impact of interventions for SpA, including axSpA. The 17-item instrument has scores ranging from 0 (good health) to 17 (poor health). Each item consists of one question that the participant needs to respond to with either "I agree" (score of 1) or "I do not agree" (score of 0). A score of "1" is given where the item is affirmed, indicating adverse health. All item scores are summed to give a total score or index. LS Mean was derived MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
score on a scale | -2.57 (0.455) | -3.16 (0.395) | -3.54 (0.396)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.330, Mixed Models Analysis; LS Mean Difference = -0.59, 95% CI 2-sided [-1.77 to 0.60], Standard Error of Mean 0.601
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.110, Mixed Models Analysis; LS Mean Difference = -0.97, 95% CI 2-sided [-2.15 to 0.22], Standard Error of Mean 0.602

25. Secondary Outcome: Change From Baseline in the Jenkins Sleep Evaluation Questionnaire (JSEQ)
Description: Jenkins Sleep Evaluation Questionnaire (JSEQ) is a 4 item scale designed to estimate sleep problems in clinical research. The JSEQ assesses the frequency of sleep disturbance in 4 categories: 1) trouble falling asleep, 2) waking up several times during the night, 3) having trouble staying asleep (including waking up far too early), and 4) waking up after the usual amount of sleep feeling tired and worn out. Patients report the numbers of days they experience each of these problems in the past month on a 6 point Likert Scale ranging from 0 = "no days" to 5 = "22-30 days. The total JSEQ score ranges from 0 to 20, with higher scores indicating greater sleep disturbance. LS Mean was derived from using MMRM with treatment, geographic region, screening MRI/CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
units on a scale | -2.9 (0.63) | -3.6 (0.52) | -3.6 (0.53)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Test type: Superiority; p = 0.348, Mixed Models Analysis; LS Mean Difference = -0.8, 95% CI 2-sided [-2.4 to 0.8], Standard Error of Mean 0.81
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Test type: Superiority; p = 0.386, Mixed Models Analysis; LS Mean Difference = -0.7, 95% CI 2-sided [-2.3 to 0.9], Standard Error of Mean 0.82

26. Secondary Outcome: Change From Baseline in the Work Productivity Activity Impairment Spondyloarthritis (WPAI-SpA) Scores
Description: The WPAI-SpA consists of 6 questions to determine employment status, hours missed from work because of SpA, hours missed from work for other reasons, hours actually worked, the degree to which SpA affected work productivity while at work, and the degree to which SpA affected activities outside of work. The WPAI-SpA has been validated in the rad-axSpA patient population. Four scores are derived: percentage of absenteeism, percentage of presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism, and percentage of impairment in activities performed outside of work. The computed percentage range for each sub-scale was from 0-100, with higher scores indicating greater impairment and less productivity. LS Mean was derived from ANCOVA with treatment, geographic region, screening MRI/CRP status and baseline value.
Time Frame: Baseline, Week 52
Population: All randomized participants. For inadequate responders who were treated with open label ixekizumab 80 mg Q2W, only data up to the time of initiation of open label of ixekizumab 80 mg Q2W were included. Missing data were imputed using the modified baseline observation carried forward (mBOCF).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 105 | 96 | 102
score on a scale
  Overall Impairment Score | -13.20 (3.386) | -26.96 (3.439) | -19.49 (3.221)
  Percentage of absenteeism | -3.11 (2.215) | -9.01 (2.257) | -7.26 (2.151)
  Percentage of presenteeism | -12.40 (3.200) | -26.01 (3.245) | -18.61 (3.047)
  Percentage of impairment in activities | -14.42 (2.584) | -25.05 (2.617) | -24.41 (2.567)
Statistical Analysis 1: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Overall Impairment Score; Test type: Superiority; p = 0.005, ANCOVA; LS Mean Difference = -13.76, 95% CI 2-sided [-23.32 to -4.20], Standard Error of Mean 4.835
Statistical Analysis 2: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Overall Impairment Score; Test type: Superiority; p = 0.183, ANCOVA; LS Mean Difference = -6.29, 95% CI 2-sided [-15.58 to 3.00], Standard Error of Mean 4.697
Statistical Analysis 3: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Percentage of absenteeism; Test type: Superiority; p = 0.060, ANCOVA; LS Mean Difference = -5.90, 95% CI 2-sided [-12.05 to 0.26], Standard Error of Mean 3.114
Statistical Analysis 4: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Percentage of absenteeism; Test type: Superiority; p = 0.182, ANCOVA; LS Mean Difference = -4.15, 95% CI 2-sided [-10.27 to 1.97], Standard Error of Mean 3.098
Statistical Analysis 5: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Percentage of presentism; Test type: Superiority; p = 0.003, ANCOVA; LS Mean Difference = -13.61, 95% CI 2-sided [-22.62 to -4.60], Standard Error of Mean 4.558
Statistical Analysis 6: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Percentage of presentism; Test type: Superiority; p = 0.164, ANCOVA; LS Mean Difference = -6.21, 95% CI 2-sided [-15.00 to 2.58], Standard Error of Mean 4.446
Statistical Analysis 7: Comparison: Placebo vs Ixekizumab 80 mg Q4W; Percentage of Impairment in Activities Performed Outside of Work; Test type: Superiority; p = 0.004, LS Mean Difference; LS Mean Difference = -10.63, 95% CI 2-sided [-17.85 to -3.41], Standard Error of Mean 3.669
Statistical Analysis 8: Comparison: Placebo vs Ixekizumab 80 mg Q2W; Percentage of Impairment in Activities Performed Outside of Work; Test type: Superiority; p = 0.006, ANCOVA; LS Mean Difference = -9.99, 95% CI 2-sided [-17.12 to -2.86], Standard Error of Mean 3.621

27. Secondary Outcome: Change From Baseline in ASAS-Nonsteroidal Anti-Inflammatory Drug (NSAID) Score
Description: ASAS-NSAID score is used to present the NSAID intake by considering the type of NSAID, the total dose, & the number of days taking NSAID during a period of interest (PI). For NSAID equivalent scoring system, range is from 0 to 100, the higher the score, the greater the NSAID intake. ASAS-NSAID score= (equivalent NSAID score) x (days of intake during PI) x (days per week)/(PI in days).
Time Frame: Baseline, Week 52
Population: All randomized participants who had NSAID (including COX-2 Inhibitor) intake at Baseline. For inadequate responders who were treated with open label ixekizumab 80 mg Q2W, only data up to the time of initiation of open label of ixekizumab 80 mg Q2W were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ixekizumab 80 mg Q4W: Participants received a starting dose of 80 or 160 mg of ixekizumab given SC at week 0 and placebo followed by 80 mg ixekizumab given SC every four weeks (Q4W) to week 52.
Arm/Group | Placebo | Ixekizumab 80 mg Q4W | Ixekizumab 80 mg Q2W
Number analyzed (Participants) | 96 | 81 | 95
score on a scale | -8.89 (29.986) | -7.91 (34.257) | -5.33 (20.935)

28. Secondary Outcome: Number of Participants With Treatment Emergent (TE) Anti-Ixekizumab Antibodies
Description: A treatment-emergent positive anti-drug antibody (TE-ADA+) participant will be defined as a 4-fold increase over a positive baseline antibody titer (Tier 3); or for a negative baseline titer, a participant with an increase from the baseline to a level of ≥ 1:10.
Time Frame: Week 52
Population: All randomized participant who received at least one dose of ixekizumab during the study and had an evaluable baseline sample and at least 1 evaluable post baseline sample.
Measure: Count of Participants; unit: Participants
Groups:
- Ixe80Q2W-Q2W: Participants received a starting dose of 80 ixekizumab as an SC injection at week 0 followed by 80 mg of ixe every two weeks (Q2W) week 2 to week 52.
- Ixe80Q4W-Q4W: Participants received a starting dose of 80 ixekizumab as an SC injection followed by 80 mg of ixekizumab Q4W week 4 to week 52.
- PBO-Ixe80Q2W: Participants who received placebo in double blind period and were inadequate responders switched to ixekizumab 80 mg Q2W open-label.
- Ixe80Q4W-Q2W: Participants who received ixekizumab 80 mg Q4W in double blind period and were inadequate responders switched to ixekizumab 80 mg Q2W open label.
Arm/Group | Ixe80Q2W-Q2W | Ixe80Q4W-Q4W | PBO-Ixe80Q2W | Ixe80Q4W-Q2W
Number analyzed (Participants) | 102 | 56 | 62 | 40
Participants | 14 | 5 | 8 | 2

29. Secondary Outcome: Pharmacokinetics (PK): Trough Concentration at Steady State (Ctrough ss)
Description: PK trough serum concentration samples were collected at steady state (Ctrough ss)
Time Frame: Week 52
Population: All randomized participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Groups:
- IxeQ2W (80S)/IxeQ2W: Ixekizumab was administered subcutaneously every 2 weeks with an 80 mg starting dose at week 0.
- IxeQ2W (80S)/IxeQ2W Open Label: Ixekizumab was administered every 2 weeks with an 80 mg starting dose at Week 0, then ixekizumab 80 mg Q2W open label between Week 16 and Week 52.
- IxeQ2W (160S)/IxeQ2W: Ixekizumab was administered subcutaneously every 2 weeks with an 160 mg starting dose at week 0.
- IxeQ2W (160s)/IxeQ2W Open Label: Ixekizumab was administered subcutaneously every 2 weeks with an 160 mg starting dose at week 0 then ixekizumab 80 mg Q2W open label between Week 16 and Week 52.
- IxeQ4W (80S) IxeQ4W: Ixekizumab was administered subcutaneously every 4 weeks with an 80 mg starting dose at week 0.
- IxeQ4W (80S)/IxeQ2W Open Label: Ixekizumab was administered subcutaneously every 4 weeks with an 80 mg starting dose at week 0 then ixekizumab 80 mg Q2W open label between Week 16 and Week 52.
- IxeQ4W(160S)/IxeQ4W: Ixekizumab was administered subcutaneously every 4 weeks with an 160 mg starting dose at week 0.
- IxeQ4W (160S) IxeQ2W Open Label: Ixekizumab was administered subcutaneously every 4 weeks with an 160 mg starting dose at week 0 then ixekizumab 80 mg Q2W open label between Week 16 and Week 52.
- PBO/IxeQ2W Open Label: Placebo was administered at week 0 then ixekizumab 80 mg Q2W open label between Week 16 and Week 52.
Arm/Group | IxeQ2W (80S)/IxeQ2W | IxeQ2W (80S)/IxeQ2W Open Label | IxeQ2W (160S)/IxeQ2W | IxeQ2W (160s)/IxeQ2W Open Label | IxeQ4W (80S) IxeQ4W | IxeQ4W (80S)/IxeQ2W Open Label | IxeQ4W(160S)/IxeQ4W | IxeQ4W (160S) IxeQ2W Open Label | PBO/IxeQ2W Open Label
Number analyzed (Participants) | 32 | 18 | 28 | 24 | 28 | 19 | 28 | 21 | 55
microgram/milliliter (μg/mL) | 7.88 (73) | 9.56 (60) | 10.3 (61) | 10.4 (72) | 2.88 (49) | 6.45 (124) | 3.54 (79) | 11.5 (53) | 9.25 (66)

ADVERSE EVENTS:
Time Frame: Up to 76 Weeks
Description: All randomized participants who received at least one dose of study drug during the study. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Placebo Double-Blind Period: Participants received placebo as 2 SC injections Q2W to week 52.
- Ixekizumab 80 mg Q4W Double-Blind Period: Participants received a starting dose of 80 or 160 mg of ixekizumab given SC at week 0 followed by 80 mg ixekizumab given SC every four weeks (Q4W) to week 52.
- Ixekizumab 80 mg Q2W Double-Blind Period: Participants received a starting dose of 80 or 160 mg of ixekizumab given SC at week 0 followed by 80 mg ixekizumab given SC every two weeks (Q2W) to week 52.
- PBO IR/IxeQ2W Open Label: Participants who received placebo in double blind period and were inadequate responders as determined by investigators switched to ixekizumab 80 mg Q2W open label.
- Ixe80Q4WIR/Ixe80Q2W Open Label: Participants who received ixekizumab 80 mg Q4W in double blind period and were inadequate responders as determined by investigators switched to ixekizumab 80 mg Q2W open label.
- Ixe80Q2WIR/Ixe80Q2W Open Label: Participants who received ixekizumab 80 mg Q2W in double blind period and were inadequate responders as determined by investigators continued on the same regimen of ixekizumab 80 mg Q2W open label.
- Other Biologic Open Label; Other Biologic Post Treatment Follow-Up Period: Participants who discontinued study treatment and were on other biologic therapy prior to entering Follow-up period
Arm/Group | Placebo Double-Blind Period | Ixekizumab 80 mg Q4W Double-Blind Period | Ixekizumab 80 mg Q2W Double-Blind Period | PBO IR/IxeQ2W Open Label | Ixe80Q4WIR/Ixe80Q2W Open Label | Ixe80Q2WIR/Ixe80Q2W Open Label | Other Biologic Open Label | Placebo Post Treatment Follow-Up Period | Ixekizumab 80 mg Q4W Post Treatment Follow-Up Period | Ixekizumab 80 mg Q2W Post Treatment Follow-Up Period | Other Biologic Post Treatment Follow-Up Period
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/96 | 0/102 | 0/42 | 0/40 | 0/62 | 0/5 | 0/3 | 0/5 | 0/28 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/104 | 2/96 | 1/102 | 1/42 | 0/40 | 2/62 | 0/5 | 0/3 | 0/5 | 1/28 | 0/5
Other Adverse Events (participants affected / at risk) | 31/104 | 43/96 | 47/102 | 13/42 | 15/40 | 26/62 | 3/5 | 1/3 | 1/5 | 1/28 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Double-Blind Period (N=104) | Ixekizumab 80 mg Q4W Double-Blind Period (N=96) | Ixekizumab 80 mg Q2W Double-Blind Period (N=102) | PBO IR/IxeQ2W Open Label (N=42) | Ixe80Q4WIR/Ixe80Q2W Open Label (N=40) | Ixe80Q2WIR/Ixe80Q2W Open Label (N=62) | Other Biologic Open Label (N=5) | Placebo Post Treatment Follow-Up Period (N=3) | Ixekizumab 80 mg Q4W Post Treatment Follow-Up Period (N=5) | Ixekizumab 80 mg Q2W Post Treatment Follow-Up Period (N=28) | Other Biologic Post Treatment Follow-Up Period (N=5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactoid reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axial spondyloarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Focal dyscognitive seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Double-Blind Period (N=104) | Ixekizumab 80 mg Q4W Double-Blind Period (N=96) | Ixekizumab 80 mg Q2W Double-Blind Period (N=102) | PBO IR/IxeQ2W Open Label (N=42) | Ixe80Q4WIR/Ixe80Q2W Open Label (N=40) | Ixe80Q2WIR/Ixe80Q2W Open Label (N=62) | Other Biologic Open Label (N=5) | Placebo Post Treatment Follow-Up Period (N=3) | Ixekizumab 80 mg Q4W Post Treatment Follow-Up Period (N=5) | Ixekizumab 80 mg Q2W Post Treatment Follow-Up Period (N=28) | Other Biologic Post Treatment Follow-Up Period (N=5)
Iritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (3) | 3 (7) | 4 (11) | 2 (5) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 4 (7) | 11 (24) | 17 (56) | 3 (11) | 3 (28) | 11 (63) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0/61 (0) | 1/46 (1) | 0/53 (0) | 0/28 (0) | 1/15 (1) | 2/41 (2) | 0/4 (0) | 0/1 (0) | 0/3 (0) | 0/19 (0) | 0/4 (0)
Bronchitis (Infections and infestations) | 3 (4) | 7 (7) | 2 (2) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (11) | 18 (26) | 16 (27) | 2 (3) | 7 (10) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (4) | 4 (5) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4) | 6 (7) | 2 (2) | 3 (4) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/61 (0) | 1/46 (1) | 0/53 (0) | 0/28 (0) | 1/15 (1) | 0/41 (0) | 0/4 (0) | 0/1 (0) | 0/3 (0) | 0/19 (0) | 0/4 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 7 (7) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 6 (7) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT02757352/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT02757352/SAP_001.pdf